CLINICAL TRIAL: NCT02246673
Title: A Phase 2a, Randomized, Open-Label Study to Evaluate the Pharmacodynamic Effects and Safety of RDEA3170 Administered in Combination With Febuxostat Compared to Febuxostat Administered Alone in Adult Subjects With Gout
Brief Title: RDEA3170 and Febuxostat Combination Study in Gout Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDEA3170-204
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — verinurad; Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- RDEA3170 10 mg (Experimental): Once daily (qd) with febuxostat 40mg (qd) for 7 days, and with febuxostat 80 mg (qd) for 7 days; febuxostat 40 mg (qd) only for 7 days, and febuxostat 80 mg (qd) only for 7 days.
  Interventions: Drug: RDEA3170 10 mg; Drug: Febuxostat 40 mg; Drug: Febuxostat 80 mg
- RDEA3170 15 mg (Experimental): Once daily with febuxostat 40mg (qd) for 7 days and with febuxostat 80mg (qd) for 7 days; febuxostat 40 mg (qd) only for 7 days, and febuxostat 80 mg (qd) only for 7 days.
  Interventions: Drug: RDEA3170 15 mg; Drug: RDEA3170 5 mg; Drug: Febuxostat 40 mg; Drug: Febuxostat 80 mg
- RDEA3170 5 mg (Experimental): Once daily with febuxostat 40mg (qd) for 7 days and with febuxostat 80mg (qd) for 7 days; febuxostat 40 mg (qd) only for 7 days, and febuxostat 80 mg (qd) only for 7 days.
  Interventions: Drug: Febuxostat 40 mg; Drug: Febuxostat 80 mg
- RDEA3170 2.5 mg (Experimental): Once daily with febuxostat 40mg (qd) for 7 days and with febuxostat 80mg (qd) for 7 days; febuxostat 40 mg (qd) only for 7 days, and febuxostat 80 mg (qd) only for 7 days.
  Interventions: Drug: RDEA3170 2.5; Drug: Febuxostat 40 mg; Drug: Febuxostat 80 mg

INTERVENTIONS:
Drug: RDEA3170 15 mg
  Arms: RDEA3170 15 mg
Drug: RDEA3170 10 mg
  Arms: RDEA3170 10 mg
Drug: RDEA3170 2.5
  Arms: RDEA3170 2.5 mg
Drug: RDEA3170 5 mg
  Arms: RDEA3170 15 mg
Drug: Febuxostat 40 mg
Drug: Febuxostat 80 mg

SUMMARY:
This is a Phase 2a, randomized, open-label, multicenter study to assess the pharmacodynamic (PD) effects and safety of RDEA3170 administered in combination with febuxostat compared to febuxostat administered alone in adult subjects with gout.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study procedures and the risks involved and is willing to provide written informed consent before the first study-related activity.
* Meets one or more criteria for the diagnosis of gout as per the American Rheumatism Association Criteria for the Classification of Acute Arthritis of Primary Gout.
* Body weight ≥ 50 kg (110 lbs) and a body mass index ≥ 18 and ≤ 45 kg/m2.
* Screening serum urate level ≥ 8 mg/dL.
* Free of any clinically significant disease or medical condition, per the Investigator's judgment.

Exclusion Criteria:

* Unable to take colchicine for gout flare prophylaxis.
* History or suspicion of kidney stones.
* Any gastrointestinal disorder that affects motility and/or absorption.
* Unstable angina, New York Heart Association class III or IV heart failure, ischemic heart disease, stroke, or deep venous thrombosis within 12 months prior to Day 1; or subject is currently receiving anticoagulants.
* Screening laboratory parameters that are outside the normal limits and are considered clinically significant by the Investigator.
* Estimated creatinine clearance < 60 mL/min calculated by the Cockcroft-Gault formula using ideal body weight during the Screening period.
* Taking losartan, fenofibrate, guaifenesin, or sodium-glucose linked transporter-2 inhibitors; chronic and stable doses are permitted if doses are stable for at least 14 days prior to study medication dosing.
* Unable or unwilling to comply with the study requirements or has a situation or condition that, in the opinion of the Investigator, may interfere with participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Hall, Study Director — Ardea Biosciences, Inc.
Locations (5):
- United States (5):
  - Anaheim, California
  - Glendale, California
  - South Miami, Florida
  - Overland Park, Kansas
  - Dallas, Texas

REFERENCES:
- [Derived] Rekic D, Johansson S, Leander J. Higher Febuxostat Exposure Observed in Asian Compared with Caucasian Subjects Independent of Bodyweight. Clin Pharmacokinet. 2021 Mar;60(3):319-328. doi: 10.1007/s40262-020-00943-6. Epub 2020 Sep 19. PMID 32951150
- [Derived] Fleischmann R, Winkle P, Hall J, Valdez S, Liu S, Yan X, Hicks L, Lee C, Miner JN, Gillen M, Hernandez-Illas M. Pharmacodynamic and pharmacokinetic effects and safety of verinurad in combination with febuxostat in adults with gout: a phase IIa, open-label study. RMD Open. 2018 Apr 9;4(1):e000647. doi: 10.1136/rmdopen-2018-000647. eCollection 2018. PMID 29657831

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-four subjects were randomized and received at least 1 dose of randomized study medication. Five cohorts of approximately 12 adult subjects with gout per cohort were randomized into the study. Overall, a total of 60 subjects completed the study in accordance with the protocol.
Pre-assignment Details: Cohorts 1 through 4 were conducted sequentially and Cohort 5 was conducted following review of the available PD/PK results of Cohort 2. Subjects in Cohorts 1 through 4 were randomized to 1 of 2 treatment sequences (ABCD or DCBA) in a 1:1 ration and subjects in Cohort 5 were randomized to 1 of 2 treatment sequences (EHGF or GFHE) in a 1:1 ratio.
Groups:
- Cohort 1: (RDEA3170 10 mg + Febuxostat 40 mg; RDEA3170 10 mg + Febuxostat 80 mg)
- Cohort 2: (RDEA3170 15 mg + Febuxostat 40 mg; RDEA3170 15 mg + Febuxostat 80 mg)
- Cohort 3: (RDEA3170 5 mg + Febuxostat 40 mg; RDEA3170 5 mg + Febuxostat 80 mg)
- Cohort 4: (RDEA3170 2.5 mg + Febuxostat 40 mg; RDEA3170 2.5 mg + Febuxostat 80 mg)
- Cohort 5: (RDEA3170 10 mg + Febuxostat 40 mg; RDEA3170 15 mg + Febuxostat 40 mg; RDEA3170 20 mg + Febuxostat 40 mg)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 14 | 12 | 12 | 14 | 12
Completed | 13 | 12 | 12 | 12 | 11
Not Completed | 1 | 0 | 0 | 2 | 1
Not completed — Sponsor Decision | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 14 | 12 | 12 | 14 | 12 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45 (8.9) | 50 (8.2) | 50 (8.5) | 48 (11.5) | 49 (10.9) | 48 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 14 | 12 | 12 | 14 | 12 | 64

OUTCOME MEASURES:

1. Primary Outcome: Serum Urate Maximum Percentage (%) Change (Emax, CB)
Description: Maximum observed percentage (%) change from baseline in serum urate concentrations.
Time Frame: 28 days
Measure: Mean (Standard Error); unit: Percentage (%)
Groups:
- Febuxostat 40 mg: Days 7/14/21/28 Overall (Cohorts 1 through 5)
- Febuxostat 80 mg: Days 7/28 Overall (Cohorts 1 through 5)
- RDEA3170 10 mg + Febuxostat 40 mg: Days 7/14/21/28 Overall (Cohorts 1 and 5)
- RDEA3170 10 mg + Febuxostat 80 mg: Days 14/21 Overall (Cohort 1)
- RDEA3170 15 mg + Febuxostat 40 mg: Days 7/14/21/28 Overall (Cohorts 2 and 5)
- RDEA3170 15 mg + Febuxostat 80 mg: Days 14/21 Overall (Cohort 2)
- RDEA3170 5 mg + Febuxostat 40 mg; RDEA3170 5 mg + Febuxostat 80 mg: Days 14/21 Overall (Cohort 3)
- RDEA3170 2.5 mg + Febuxostat 40 mg; RDEA3170 2.5 mg + Febuxostat 80 mg: Days 14/21 Overall (Cohort 4)
- RDEA3170 20 mg + Febuxostat 40 mg: Days 14/21 Overall (Cohort 5)
Arm/Group | Febuxostat 40 mg | Febuxostat 80 mg | RDEA3170 10 mg + Febuxostat 40 mg | RDEA3170 10 mg + Febuxostat 80 mg | RDEA3170 15 mg + Febuxostat 40 mg | RDEA3170 15 mg + Febuxostat 80 mg | RDEA3170 5 mg + Febuxostat 40 mg | RDEA3170 5 mg + Febuxostat 80 mg | RDEA3170 2.5 mg + Febuxostat 40 mg | RDEA3170 2.5 mg + Febuxostat 80 mg | RDEA3170 20 mg + Febuxostat 40 mg
Number analyzed (Participants) | 58 | 47 | 22 | 10 | 23 | 11 | 12 | 12 | 12 | 12 | 11
Percentage (%) | -43.5 (1.10) | -55.6 (1.37) | -70.4 (1.35) | -79.1 (2.53) | -74.9 (1.18) | -82.4 (1.76) | -59.4 (2.81) | -66.7 (2.32) | -52.5 (2.51) | -62.7 (2.69) | -77.3 (1.18)
Statistical Analysis 1: Comparison: Febuxostat 40 mg vs RDEA3170 10 mg + Febuxostat 40 mg; Cohort 1; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = -28.18, 95% CI 2-sided [-33.85 to -22.51]
Statistical Analysis 2: Comparison: Febuxostat 80 mg vs RDEA3170 10 mg + Febuxostat 80 mg; Cohort 1; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = -25.29, 95% CI 2-sided [-31.23 to -19.34]
Statistical Analysis 3: Comparison: Febuxostat 40 mg vs RDEA3170 15 mg + Febuxostat 40 mg; Cohort 2; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = -29.15, 95% CI 2-sided [-33.15 to -25.15]
Statistical Analysis 4: Comparison: Febuxostat 80 mg vs RDEA3170 15 mg + Febuxostat 80 mg; Cohort 2; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = -22.25, 95% CI 2-sided [-26.36 to -18.14]
Statistical Analysis 5: Comparison: Febuxostat 40 mg vs RDEA3170 5 mg + Febuxostat 40 mg; Cohort 3; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = -17.52, 95% CI 2-sided [-21.54 to -13.50]
Statistical Analysis 6: Comparison: Febuxostat 80 mg vs RDEA3170 5 mg + Febuxostat 80 mg; Cohort 3; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = -15.51, 95% CI 2-sided [-19.53 to -11.49]
Statistical Analysis 7: Comparison: Febuxostat 40 mg vs RDEA3170 2.5 mg + Febuxostat 40 mg; Cohort 4; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = -9.74, 95% CI 2-sided [-13.97 to -5.51]
Statistical Analysis 8: Comparison: Febuxostat 80 mg vs RDEA3170 2.5 mg + Febuxostat 80 mg; Cohort 4; Test type: Superiority or Other; p = 0.0221, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = -4.98, 95% CI 2-sided [-9.19 to -0.76]
Statistical Analysis 9: Comparison: Febuxostat 40 mg vs RDEA3170 20 mg + Febuxostat 40 mg; Cohort 5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = -35.38, 95% CI 2-sided [-38.89 to -31.87]
Statistical Analysis 10: Comparison: Febuxostat 40 mg vs RDEA3170 10 mg + Febuxostat 40 mg; Cohort 5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = -27.08, 95% CI 2-sided [-30.60 to -23.57]
Statistical Analysis 11: Comparison: Febuxostat 40 mg vs RDEA3170 15 mg + Febuxostat 40 mg; Cohort 5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = -31.26, 95% CI 2-sided [-34.77 to -27.75]

2. Primary Outcome: Urine Uric Acid % Change (0-24h) (Aeur, CB)
Description: Percentage (%) change from baseline in the amount of uric acid recovered in urine.
Time Frame: 28 days
Measure: Mean (Standard Error); unit: Percentage (%)
Groups:
- Febuxostat 80 mg: Days 14/21 Overall (Cohorts 1 through 5)
Arm/Group | Febuxostat 40 mg | Febuxostat 80 mg | RDEA3170 10 mg + Febuxostat 40 mg | RDEA3170 10 mg + Febuxostat 80 mg | RDEA3170 15 mg + Febuxostat 40 mg | RDEA3170 15 mg + Febuxostat 80 mg | RDEA3170 5 mg + Febuxostat 40 mg | RDEA3170 5 mg + Febuxostat 80 mg | RDEA3170 2.5 mg + Febuxostat 40 mg | RDEA3170 2.5 mg + Febuxostat 80 mg | RDEA3170 20 mg + Febuxostat 40 mg
Number analyzed (Participants) | 56 | 45 | 24 | 13 | 22 | 10 | 10 | 10 | 11 | 11 | 10
Percentage (%) | -48.6 (1.71) | -60.3 (1.58) | -23.7 (5.56) | -36.6 (6.75) | -22.9 (4.15) | -44.4 (5.57) | -26.2 (8.28) | -39.2 (5.95) | -40.2 (4.07) | -61.1 (2.16) | -14.2 (10.9)
Statistical Analysis 1: Comparison: Febuxostat 40 mg vs RDEA3170 10 mg + Febuxostat 40 mg; Cohort 1; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 24.27, 95% CI 2-sided [12.57 to 35.98]
Statistical Analysis 2: Comparison: Febuxostat 80 mg vs RDEA3170 10 mg + Febuxostat 80 mg; Cohort 1; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 20.08, 95% CI 2-sided [8.38 to 31.79]
Statistical Analysis 3: Comparison: Febuxostat 40 mg vs RDEA3170 15 mg + Febuxostat 40 mg; Cohort 2; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 23.70, 95% CI 2-sided [14.23 to 33.17]
Statistical Analysis 4: Comparison: Febuxostat 80 mg vs RDEA3170 15 mg + Febuxostat 80 mg; Cohort 2; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 18.37, 95% CI 2-sided [8.30 to 28.44]
Statistical Analysis 5: Comparison: Febuxostat 40 mg vs RDEA3170 5 mg + Febuxostat 40 mg; Cohort 3; Test type: Superiority or Other; p = 0.0101, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 18.82, 95% CI 2-sided [4.86 to 32.79]
Statistical Analysis 6: Comparison: Febuxostat 80 mg vs RDEA3170 5 mg + Febuxostat 80 mg; Cohort 3; Test type: Superiority or Other; p = 0.0055, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 20.52, 95% CI 2-sided [6.56 to 34.48]
Statistical Analysis 7: Comparison: Febuxostat 40 mg vs RDEA3170 2.5 mg + Febuxostat 40 mg; Cohort 4; Test type: Superiority or Other; p = 0.0065, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 10.36, 95% CI 2-sided [3.13 to 17.59]
Statistical Analysis 8: Comparison: Febuxostat 80 mg vs RDEA3170 2.5 mg + Febuxostat 80 mg; Cohort 4; Test type: Superiority or Other; p = 0.6140, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 1.79, 95% CI 2-sided [-5.37 to 8.94]
Statistical Analysis 9: Comparison: Febuxostat 40 mg vs RDEA3170 20 mg + Febuxostat 40 mg; Cohort 5; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 30.83, 95% CI 2-sided [15.62 to 46.04]
Statistical Analysis 10: Comparison: Febuxostat 40 mg vs RDEA3170 10 mg + Febuxostat 40 mg; Cohort 5; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 24.38, 95% CI 2-sided [9.63 to 39.14]
Statistical Analysis 11: Comparison: Febuxostat 40 mg vs RDEA3170 15 mg + Febuxostat 40 mg; Cohort 5; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 26.35, 95% CI 2-sided [11.59 to 41.11]

3. Primary Outcome: Renal Clearance of Uric Acid % Change (0-24h) (CLur, CB)
Description: Percentage (%) change from baseline in renal clearance of uric acid.
Time Frame: 28 days
Measure: Mean (Standard Error); unit: Percentage (%)
Arm/Group | Febuxostat 40 mg | Febuxostat 80 mg | RDEA3170 10 mg + Febuxostat 40 mg | RDEA3170 10 mg + Febuxostat 80 mg | RDEA3170 15 mg + Febuxostat 40 mg | RDEA3170 15 mg + Febuxostat 80 mg | RDEA3170 5 mg + Febuxostat 40 mg | RDEA3170 5 mg + Febuxostat 80 mg | RDEA3170 2.5 mg + Febuxostat 40 mg | RDEA3170 2.5 mg + Febuxostat 80 mg | RDEA3170 20 mg + Febuxostat 40 mg
Number analyzed (Participants) | 50 | 37 | 21 | 10 | 20 | 10 | 10 | 10 | 10 | 10 | 9
Percentage (%) | -15.2 (2.53) | -18.8 (2.52) | 125 (17.4) | 153 (30.5) | 157 (15.9) | 172 (30.0) | 58.7 (15.7) | 68.4 (24.7) | 20.9 (10.1) | 0.011 (7.36) | 223 (47.0)
Statistical Analysis 1: Comparison: Febuxostat 40 mg vs RDEA3170 10 mg + Febuxostat 40 mg; Cohort 1; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 139.11, 95% CI 2-sided [93.92 to 184.31]
Statistical Analysis 2: Comparison: Febuxostat 80 mg vs RDEA3170 10 mg + Febuxostat 80 mg; Cohort 1; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 174.47, 95% CI 2-sided [125.52 to 233.42]
Statistical Analysis 3: Comparison: Febuxostat 40 mg vs RDEA3170 15 mg + Febuxostat 40 mg; Cohort 2; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 168.03, 95% CI 2-sided [123.13 to 212.93]
Statistical Analysis 4: Comparison: Febuxostat 80 mg vs RDEA3170 15 mg + Febuxostat 80 mg; Cohort 2; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 188.75, 95% CI 2-sided [138.04 to 239.46]
Statistical Analysis 5: Comparison: Febuxostat 40 mg vs RDEA3170 5 mg + Febuxostat 40 mg; Cohort 3; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 70.43, 95% CI 2-sided [33.74 to 107.12]
Statistical Analysis 6: Comparison: Febuxostat 80 mg vs RDEA3170 5 mg + Febuxostat 80 mg; Cohort 3; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 91.50, 95% CI 2-sided [54.81 to 128.19]
Statistical Analysis 7: Comparison: Febuxostat 40 mg vs RDEA3170 2.5 mg + Febuxostat 40 mg; Cohort 4; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 40.11, 95% CI 2-sided [25.17 to 55.05]
Statistical Analysis 8: Comparison: Febuxostat 80 mg vs RDEA3170 2.5 mg + Febuxostat 80 mg; Cohort 4; Test type: Superiority or Other; p = 0.0350, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 15.96, 95% CI 2-sided [1.20 to 30.71]
Statistical Analysis 9: Comparison: Febuxostat 40 mg vs RDEA3170 20 mg + Febuxostat 40 mg; Cohort 5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 236.08, 95% CI 2-sided [178.29 to 293.86]
Statistical Analysis 10: Comparison: Febuxostat 40 mg vs RDEA3170 10 mg + Febuxostat 40 mg; Cohort 5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 146.20, 95% CI 2-sided [90.40 to 202.01]
Statistical Analysis 11: Comparison: Febuxostat 40 mg vs RDEA3170 15 mg + Febuxostat 40 mg; Cohort 5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 176.57, 95% CI 2-sided [120.77 to 232.38]

4. Primary Outcome: Fract. Excretion of Uric Acid % Change (0-24h) (FEUA, CB)
Description: Percentage (%) change from baseline in fractional excretion of uric acid.
Time Frame: 28 days
Measure: Mean (Standard Error); unit: Percentage (%)
Arm/Group | Febuxostat 40 mg | Febuxostat 80 mg | RDEA3170 10 mg + Febuxostat 40 mg | RDEA3170 10 mg + Febuxostat 80 mg | RDEA3170 15 mg + Febuxostat 40 mg | RDEA3170 15 mg + Febuxostat 80 mg | RDEA3170 5 mg + Febuxostat 40 mg | RDEA3170 5 mg + Febuxostat 80 mg | RDEA3170 2.5 mg + Febuxostat 40 mg | RDEA3170 2.5 mg + Febuxostat 80 mg | RDEA3170 20 mg + Febuxostat 40 mg
Number analyzed (Participants) | 47 | 33 | 21 | 8 | 19 | 10 | 7 | 7 | 10 | 10 | 9
Percentage (%) | -20.6 (1.82) | -20.8 (2.62) | 100 (13.4) | 155 (32.4) | 133 (12.2) | 152 (26.2) | 46.6 (9.36) | 54.8 (20.5) | 15.2 (9.30) | 4.73 (6.15) | 162 (23.2)
Statistical Analysis 1: Comparison: Febuxostat 40 mg vs RDEA3170 10 mg + Febuxostat 40 mg; Cohort 1; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 135.82, 95% CI 2-sided [93.33 to 178.32]
Statistical Analysis 2: Comparison: Febuxostat 80 mg vs RDEA3170 10 mg + Febuxostat 80 mg; Cohort 1; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 178.58, 95% CI 2-sided [129.25 to 227.90]
Statistical Analysis 3: Comparison: Febuxostat 40 mg vs RDEA3170 15 mg + Febuxostat 40 mg; Cohort 2; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 163.98, 95% CI 2-sided [120.80 to 207.16]
Statistical Analysis 4: Comparison: Febuxostat 80 mg vs RDEA3170 15 mg + Febuxostat 80 mg; Cohort 2; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 169.93, 95% CI 2-sided [122.82 to 217.03]
Statistical Analysis 5: Comparison: Febuxostat 40 mg vs RDEA3170 5 mg + Febuxostat 40 mg; Cohort 3; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 59.60, 95% CI 2-sided [28.85 to 90.34]
Statistical Analysis 6: Comparison: Febuxostat 80 mg vs RDEA3170 5 mg + Febuxostat 80 mg; Cohort 3; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 73.54, 95% CI 2-sided [42.79 to 104.28]
Statistical Analysis 7: Comparison: Febuxostat 40 mg vs RDEA3170 2.5 mg + Febuxostat 40 mg; Cohort 4; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 33.70, 95% CI 2-sided [21.21 to 46.20]
Statistical Analysis 8: Comparison: Febuxostat 80 mg vs RDEA3170 2.5 mg + Febuxostat 80 mg; Cohort 4; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 27.08, 95% CI 2-sided [14.58 to 39.58]
Statistical Analysis 9: Comparison: Febuxostat 40 mg vs RDEA3170 20 mg + Febuxostat 40 mg; Cohort 5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 188.83, 95% CI 2-sided [152.55 to 225.10]
Statistical Analysis 10: Comparison: Febuxostat 40 mg vs RDEA3170 10 mg + Febuxostat 40 mg; Cohort 5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 116.83, 95% CI 2-sided [81.76 to 151.90]
Statistical Analysis 11: Comparison: Febuxostat 40 mg vs RDEA3170 15 mg + Febuxostat 40 mg; Cohort 5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The model included treatment and period as fixed effects and subject(s) as a random effect; Geometric Least Squares mean Ratio = 151.66, 95% CI 2-sided [116.59 to 186.73]

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax of multiple-dose RDEA3170 administered in combination with febuxostat from plasma
Time Frame: Days 7 to 28
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- RDEA3170 10 mg + Febuxostat 40 mg: Overall (Cohorts 1 and 5)
- RDEA3170 10 mg + Febuxostat 80 mg: Overall (Cohort 1)
- RDEA3170 15 mg + Febuxostat 40 mg: Overall (Cohorts 2 and 5)
- RDEA3170 15 mg + Febuxostat 80 mg: Overall (Cohort 2)
- RDEA3170 5 mg + Febuxostat 40 mg; RDEA3170 5 mg + Febuxostat 80 mg: Overall (Cohort 3)
- RDEA3170 2.5 mg + Febuxostat 40 mg; RDEA3170 2.5 mg + Febuxostat 80 mg: Overall (Cohort 4)
- RDEA3170 20 mg + Febuxostat 40 mg: Overall (Cohort 5)
Arm/Group | RDEA3170 10 mg + Febuxostat 40 mg | RDEA3170 10 mg + Febuxostat 80 mg | RDEA3170 15 mg + Febuxostat 40 mg | RDEA3170 15 mg + Febuxostat 80 mg | RDEA3170 5 mg + Febuxostat 40 mg | RDEA3170 5 mg + Febuxostat 80 mg | RDEA3170 2.5 mg + Febuxostat 40 mg | RDEA3170 2.5 mg + Febuxostat 80 mg | RDEA3170 20 mg + Febuxostat 40 mg
Number analyzed (Participants) | 24 | 13 | 23 | 11 | 12 | 12 | 12 | 12 | 11
ng/mL | 15.5 [12.9 to 18.6] | 16.1 [12.6 to 20.6] | 21.2 [18.0 to 25.1] | 20.4 [15.8 to 26.2] | 7.20 [5.55 to 9.34] | 7.54 [5.69 to 9.99] | 3.45 [2.63 to 4.52] | 3.37 [2.42 to 4.68] | 26.1 [20.1 to 33.9]

6. Secondary Outcome: Time of Occurrence of Maximum Observed Concentration (Tmax)
Description: Tmax of multiple-dose RDEA3170 administered in combination with febuxostat from plasma
Time Frame: Days 7 to 28
Measure: Median (Full Range); unit: hr
Arm/Group | RDEA3170 10 mg + Febuxostat 40 mg | RDEA3170 10 mg + Febuxostat 80 mg | RDEA3170 15 mg + Febuxostat 40 mg | RDEA3170 15 mg + Febuxostat 80 mg | RDEA3170 5 mg + Febuxostat 40 mg | RDEA3170 5 mg + Febuxostat 80 mg | RDEA3170 2.5 mg + Febuxostat 40 mg | RDEA3170 2.5 mg + Febuxostat 80 mg | RDEA3170 20 mg + Febuxostat 40 mg
Number analyzed (Participants) | 24 | 13 | 23 | 11 | 12 | 12 | 12 | 12 | 11
hr | 3.00 [1.50 to 10.0] | 3.00 [1.00 to 12.0] | 3.00 [1.50 to 8.00] | 4.00 [2.00 to 6.00] | 3.50 [2.00 to 6.00] | 4.00 [1.50 to 12.0] | 3.50 [1.50 to 8.00] | 2.50 [1.00 to 10.0] | 3.00 [1.50 to 6.00]

7. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero up to 24 Hours Postdose (AUC 0-24)
Description: AUC 0-24 of multiple-dose RDEA3170 administered in combination with febuxostat from plasma
Time Frame: Days 7 to 28
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | RDEA3170 10 mg + Febuxostat 40 mg | RDEA3170 10 mg + Febuxostat 80 mg | RDEA3170 15 mg + Febuxostat 40 mg | RDEA3170 15 mg + Febuxostat 80 mg | RDEA3170 5 mg + Febuxostat 40 mg | RDEA3170 5 mg + Febuxostat 80 mg | RDEA3170 2.5 mg + Febuxostat 40 mg | RDEA3170 2.5 mg + Febuxostat 80 mg | RDEA3170 20 mg + Febuxostat 40 mg
Number analyzed (Participants) | 24 | 13 | 23 | 11 | 12 | 12 | 12 | 12 | 11
ng·hr/mL | 123 [104 to 146] | 138 [106 to 179] | 186 [164 to 212] | 225 [182 to 278] | 62.2 [47.8 to 80.8] | 57.6 [46.8 to 70.9] | 28.0 [21.2 to 36.9] | 27.4 [19.7 to 38.1] | 216 [173 to 270]

8. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Sampling Timepoint (AUC Last)
Description: AUC last of multiple-dose RDEA3170 administered in combination with febuxostat from plasma
Time Frame: Days 7 to 28
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | RDEA3170 10 mg + Febuxostat 40 mg | RDEA3170 10 mg + Febuxostat 80 mg | RDEA3170 15 mg + Febuxostat 40 mg | RDEA3170 15 mg + Febuxostat 80 mg | RDEA3170 5 mg + Febuxostat 40 mg | RDEA3170 5 mg + Febuxostat 80 mg | RDEA3170 2.5 mg + Febuxostat 40 mg | RDEA3170 2.5 mg + Febuxostat 80 mg | RDEA3170 20 mg + Febuxostat 40 mg
Number analyzed (Participants) | 24 | 13 | 23 | 11 | 12 | 12 | 12 | 12 | 11
ng·hr/mL | 123 [104 to 146] | 138 [106 to 179] | 186 [164 to 212] | 225 [182 to 278] | 62.2 [47.8 to 80.8] | 62.6 [48.2 to 81.3] | 28.0 [21.2 to 36.9] | 26.8 [18.8 to 38.3] | 216 [173 to 270]

9. Secondary Outcome: Apparent Terminal Half-life (t1/2)
Description: t1/2 of multiple-dose RDEA3170 administered in combination with febuxostat from plasma
Time Frame: Days 7 to 28
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | RDEA3170 10 mg + Febuxostat 40 mg | RDEA3170 10 mg + Febuxostat 80 mg | RDEA3170 15 mg + Febuxostat 40 mg | RDEA3170 15 mg + Febuxostat 80 mg | RDEA3170 5 mg + Febuxostat 40 mg | RDEA3170 5 mg + Febuxostat 80 mg | RDEA3170 2.5 mg + Febuxostat 40 mg | RDEA3170 2.5 mg + Febuxostat 80 mg | RDEA3170 20 mg + Febuxostat 40 mg
Number analyzed (Participants) | 24 | 12 | 23 | 11 | 12 | 11 | 12 | 12 | 11
hr | 8.26 [6.71 to 10.2] | 9.64 [6.77 to 13.7] | 10.6 [8.41 to 13.3] | 10.8 [8.17 to 14.3] | 13.2 [8.11 to 21.4] | 11.3 [7.09 to 18.1] | 13.0 [8.89 to 19.1] | 12.5 [8.18 to 19.2] | 11.6 [7.17 to 18.8]

10. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Time Frame: 10 weeks
Measure: Number; unit: Number of participants
Groups:
- Febuxostat 40 mg; Febuxostat 80 mg: Overall (Cohorts 1 through 5)
Arm/Group | Febuxostat 40 mg | Febuxostat 80 mg | RDEA3170 10 mg + Febuxostat 40 mg | RDEA3170 10 mg + Febuxostat 80 mg | RDEA3170 15 mg + Febuxostat 40 mg | RDEA3170 15 mg + Febuxostat 80 mg | RDEA3170 5 mg + Febuxostat 40 mg | RDEA3170 5 mg + Febuxostat 80 mg | RDEA3170 2.5 mg + Febuxostat 40 mg | RDEA3170 2.5 mg + Febuxostat 80 mg | RDEA3170 20 mg + Febuxostat 40 mg
Number analyzed (Participants) | 61 | 51 | 25 | 13 | 23 | 12 | 12 | 12 | 12 | 13 | 11
Number of participants | 3 | 8 | 4 | 6 | 1 | 0 | 0 | 1 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Febuxostat 40 mg | Febuxostat 80 mg | Overall RDEA3170 + Febuxostat Combination
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/51 | 0/62
Other Adverse Events (participants affected / at risk) | 3/61 | 8/51 | 13/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Febuxostat 40 mg (N=61) | Febuxostat 80 mg (N=51) | Overall RDEA3170 + Febuxostat Combination (N=62)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Aphthous Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes Simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tympanic Membrane Hyperaemia (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.